CLINICAL TRIAL: NCT04529928
Title: An Initial Evaluation of the Carillon Mitral Contour System for Treatment of Atrial Function Mitral Regurgitation
Acronym: AFIRE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not accruing subjects as expected, due to limits in hospital resources and staff as a result of the COVID pandemic in Europe.
Sponsor: Cardiac Dimensions Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVP-3473-01
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Functional Mitral Regurgitation; Atrial Fibrillation; Atrial Functional Mitral Regurgitation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implanted (Experimental): Subjects successfully implanted with the Carillon Mitral Contour System
  Interventions: Device: Carillon Mitral Contour System

INTERVENTIONS:
Device: Carillon Mitral Contour System — Eligible subjects will be implanted with the Carillon Device, utilizing the Carillon Mitral Contour System. The device is a permanent implant in the coronary sinus/great cardiac vein, designed to cinch the mitral annulus. The implant procedure is minimally invasive, conducted via catheter placement.
  Other Names: Carillon; Carillon Device; Carillon Implant

SUMMARY:
The objective of this prospective, multi-center trial is to assess the effectiveness of the CARILLON Mitral Contour System in treating patients with moderate-to-severe atrial functional mitral regurgitation (aFMR)

DETAILED DESCRIPTION:
The AFIRE Trial is a prospective, multi-center clinical trial.

The centers will utilize pre-screening of existing medical records to identify potentially eligible subjects. Once informed consent has been obtained, the subject will undergo baseline assessments, which include: Transthoracic echocardiography, transesophageal echocardiography, and functional assessments (Six-Minute Walk Test, NYHA, and Quality of Life Questionnaires). Following final eligibility determination, eligible subjects will under the index procedure to implant the Carillon device (includes coronary sinus venogram). Subject will be discharged following one-night in-hospital stay and discharge assessments.

Subjects who have the Carillon implant procedure attempted but were not successfully implanted (Non-Implanted subjects) will be followed through discharge or resolution of safety events, whichever is longer, and then discharged from the trial.

Implanted subjects will have follow-up assessments performed at 1 month, 6 months, and 12 months post index procedure. Follow-up assessments will include transthoracic echocardiography, Six-Minute Walk Test, and Quality of Life Questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate-to-severe non-primary Mitral Regurgitation (as assessed by qualitative, semi-quantitative and/or quantitative echocardiographic assessment in the setting of all of the following:

   a. Severe left atrial (LA) dilatation as defined by at least two (2) of the following: i. LA area ≥ 41cm2 ii. Indexed LA volume > 48mL/m2 iii. LA diameter ≥ 52 mm for men and ≥ 46 mm for women b. Preserved left ventricular contractility (Left Ventricular Ejection Fraction ≥50% by Simpson's biplane technique) c. No more than mild left ventricular dilatation as defined by: i. LV diastolic volume/BSA (mL/m2) <90 mL/m2 for men and <71 mL/m2 for women ii. LV systolic volume/BSA (mL/m2) <39 mL/m2 for men and <33 mL/m2 for women
2. New York Heart Association (NYHA) Class II, III or ambulatory IV heart failure
3. Stable heart failure medication regimen for at least 30 days prior to index procedure including antihypertensives and/or diuretics to achieve controlled BP (< 140 mmHg systolic) and adequate heart rate control (<100 bpm resting HR)
4. Patient deemed appropriate candidate for transcatheter mitral valve repair by the local multidisciplinary heart team
5. Subject meets anatomic screening criteria as determined by angiographic screening at the time of the index procedure to ensure that implant can be sized and placed in accordance with the Instructions for Use
6. Female subjects of child-bearing potential must have a negative serum BHCG test
7. Age ≥ 18 years old
8. The subject has read the informed consent, agrees to comply with the requirements, and has signed the informed consent to participate in the study

Exclusion Criteria:

1. Hospitalization in past three (3) months due to myocardial infarction, coronary artery bypass graft surgery, and/or unstable angina
2. Evidence of transient ischemic attack or stroke within three (3) months prior to intervention
3. Percutaneous coronary intervention in the last 30 days
4. Subjects expected to require any cardiac surgery, including surgery for coronary artery disease or for pulmonic, aortic, or tricuspid valve disease within one (1) year
5. Subjects expected to require any percutaneous coronary intervention within 30 days of the index procedure.
6. Pre-existing device (e.g., pacing lead) in coronary sinus (CS) / great cardiac vein (GCV), or anticipated need for cardiac resynchronization therapy (CRT) within twelve (12) months
7. Presence of a coronary artery stent under the CS / GCV in the implant target zone
8. Presence of left atrial appendage (LAA) clot.
9. Presence of primary renal dysfunction or significantly compromised renal function as reflected by a serum creatinine > 2.2 mg/dL (194.5 µmol/L) OR estimated Glomerular Filtration Rate (eGFR) < 30 ml/min
10. Poorly controlled atrial fibrillation or flutter, with poor ventricular rate control (> 100 bpm resting HR), or other poorly controlled symptomatic brady- or tachy-arrhythmias
11. Uncontrolled hypertension (BP > 180 mmHg systolic and/or >105 mmHg diastolic) or hypotension (BP < 90 mmHg systolic) at baseline
12. Presence of severe mitral annular calcification
13. Prior mitral valve surgery
14. Presence of a mechanical mitral heart valve, mitral bio-prosthetic valve or mitral annuloplasty ring
15. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
16. Active endocarditis
17. Severe aortic stenosis (aortic valve area <1.0 cm2) or severe aortic regurgitation
18. Infiltrative cardiomyopathies (e.g., amyloidosis, hemochromatosis, sarcoidosis)
19. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than atrial functional mitral regurgitation
20. Subjects with echocardiographic documentation of non-compaction cardiomyopathy with associated hypercontractility of the cardiac structures supporting the mitral annulus
21. Hemodynamic instability requiring inotropic support or mechanical heart circulatory support
22. Active infections requiring current antibiotic therapy
23. Severe right ventricular failure or severe tricuspid regurgitation
24. History of bleeding diathesis or coagulopathy, or subject who refuses blood transfusions
25. Significant organic mitral valve pathology (e.g., moderate or severe myxomatous degeneration, with or without mitral leaflet prolapse, rheumatic disease, full or partial chordal rupture)
26. Allergy to contrast dye that cannot be pre-medicated
27. Pregnant or planning pregnancy within next 12 months.
28. Chronic severe pathology limiting survival to less than 12-months in the judgement of the investigator
29. Anticipated need of left ventricular assist device within twelve (12) months
30. Currently participating or has participated in another investigational study where the study primary endpoint was not reached at the time of screening
31. Patient requires emergent/emergency treatment for mitral regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Change in mitral regurgitant volume (mL) associated with the Carillon device at 6 months post-implant, as compared to baseline | 6 Months

CONTACTS AND LOCATIONS:
Locations (2):
- Royal Prince Alfred, Sydney, New South Wales, Australia
- European Interbalkan Medical Center, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No